CLINICAL TRIAL: NCT00559962
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group Study to Evaluate Low Doses of the MTP-Inhibitor AEGR-733 on Hepatic Fat Accumulation as Measured by Magnetic Resonance Spectroscopy
Brief Title: Evaluate Low Doses of AEGR-733 on Hepatic Fat Accumulation by MRS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aegerion Pharmaceuticals, Inc. (Industry)
Responsible Party: William J Sasiela, PhD Chief Medical Officer, Aegerion Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AEGR-733-004
Record Dates: First submitted 2007-11-15; First posted 2007-11-19 (Estimated); Results first posted 2013-02-22 (Estimated); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Hyperlipidemia
Keywords: LDL; hepatic fat
MeSH Terms: conditions — Hyperlipidemias | interventions — BMS201038; Atorvastatin; Fenofibrate; Ezetimibe

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- 1 (Placebo Comparator): Placebo
  Interventions: Drug: placebo
- 2 (Active Comparator): 2.5 mg AEGR-733
  Interventions: Drug: AEGR-733
- 3 (Active Comparator): 5 mg AEGR-733
  Interventions: Drug: AEGR-733
- 4 (Active Comparator): 7.5 mg AEGR-733
  Interventions: Drug: AEGR-733
- 5 (Active Comparator): 10 mg AEGR-733
  Interventions: Drug: AEGR-733
- 6 (Active Comparator): 5 mg AEGR-733 + 20 mg atorvastatin
  Interventions: Drug: AEGR-733 and atorvastatin
- 7 (Active Comparator): 5 mg AEGR-733 + 145 mg fenofibrate
  Interventions: Drug: AEGR-733 and fenofibrate
- 8 (Active Comparator): 5 mg AEGR-733 + 10 mg ezetimibe
  Interventions: Drug: AEGR-733 and ezetimibe

INTERVENTIONS:
Drug: AEGR-733 — 3 capsules each evening for each 4-week period
  Arms: 2
Drug: placebo — 3 capsules each evening for each 4-week period
  Arms: 1
Drug: AEGR-733 — 3 capsules each evening for each 4-week period
  Arms: 3
Drug: AEGR-733 — 3 capsules each evening for each 4-week period
  Arms: 4
Drug: AEGR-733 — 3 capsules each evening for each 4-week period
  Arms: 5
Drug: AEGR-733 and atorvastatin — 3 capsules each evening for each 4-week period
  Arms: 6
Drug: AEGR-733 and fenofibrate — 3 capsules each evening for each 4-week period
  Arms: 7
Drug: AEGR-733 and ezetimibe — 3 capsules each evening for each 4-week period
  Arms: 8

SUMMARY:
To determine safety and effectiveness of low-dose therapeutic AEGR-733 +/- atorvastatin, ezetimibe or fenofibrate (compared to placebo) on liver fat accumulation measured by Magnetic Resonance Spectroscopy

DETAILED DESCRIPTION:
The goal within the current development program and this study is to investigate whether lower doses of AEGR-733 can result in significant reductions in LDL-C and TGs while providing fewer gastrointestinal adverse events and less hepatic fat accumulation than seen in studies with higher doses. The potential for atorvastatin, ezetimibe or the PPAR-alpha agonist (fenofibrate) to ameliorate any hepatic fat accumulation will also be investigated. The twelve week dosing schedule allows us to demonstrate the longer term effects of lower doses of MTP-I on hepatic fat accumulation.

ELIGIBILITY:
Inclusion Criteria:

1. LDL-C between 100 and 190 mg/dL
2. Hepatic fat under 6.2% per MRS

Exclusion Criteria:

1. Pregnant or lactating females
2. Uncontrolled hypertension >180/95 mmHg
3. Chronic renal insufficiency - serum creatinine >2.5 mg/dL at screen
4. Liver disease; i.e., hepatitis, cirrhosis
5. Major surgery within 3 months of screen
6. Cardiac insufficiency
7. Hx of malignancy other than basal or squamous cell within past 5 yrs
8. Participation in any investigational drug study within 6 wks of screen
9. Prior exposure to AEGR-733 in past 12 months
10. Serious or unstable medical or psychological conditions
11. More than one alcoholic drink per day
12. Regular consumption of grapefruit juice or meds known to be metabolized by CYP 3A4
13. Currently taking corticosteroids
14. Other lipid-lowering meds (washout permitted)
15. Fish oil, niacin grater than 200 mg/day and herbal weight loss products (washout permitted)
16. Acute CVD or event within previous 6 months
17. Diabetes Mellitus
18. Hepatitis B or C
19. Medicated COPD
20. Idiopathic pulmonary fibrosis
21. G.I. disorders that cause chronic diarrhea
22. Fasting triglycerides =/> 400 mg/dL
23. Body Mass Index > 35kg/m2

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2007-10; Primary Completion 2008-10 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Sasiela, PhD, Study Director — Aegerion Pharmaceuticals, Inc.
Locations (15):
- United States (15):
  - Scripps Clinic, San Diego, California
  - Radiant Research, Santa Rosa, California
  - MedStar Research Institute, Washington D.C., District of Columbia
  - Radiant Research, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - LMARC, Louisville, Kentucky
  - Maine Research Associates, Auburn, Maine
  - Health Trends Research, Baltimore, Maryland
  - Johns Hopkins, Baltimore, Maryland
  - Washington Univ. School of Medicine, St Louis, Missouri
  - Sterling Research Group, Cincinnati, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - Clinical Trial Network, Houston, Texas
  - dgd Research, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was performed from 06 Sept 2007 to 05 Sept 2008. A total of 16 medical clinics participated in the study.
Pre-assignment Details: Subjects underwent a 5- to 9-week screening washout period to determine study eligibility and to wash-out patients of all lipid-lowering therapies; patients were required to have low-density lipoprotein cholesterol (LDL-C) between 100 and 190 mg/dL (average of 2 visits during screening) and hepatic fat less than 6.2% for randomization.
Groups:
- Placebo: Oral placebo every 4 weeks for 12 weeks
- AEGR-733 2.5 mg: Oral lomitapide 2.5 mg every 4 weeks for 12 weeks
- AEGR-733 5 mg: Oral lomitapide 5 mg every 4 weeks for 12 weeks
- AEGR-733 7.5 mg: Oral lomitapide 7.5 mg every 4 weeks for 12 weeks
- AEGR-733 10 mg: Oral lomitapide 10 mg every 4 weeks for 12 weeks
- AEGR-733 5 mg + Atorvastatin 20 mg: Oral lomitapide 5 mg + atorvastatin 20 mg every 4 weeks for 12 weeks
- AEGR-733 5 mg + Fenofibrate 145 mg: Oral lomitapide 5 mg + micronized fenofibrate 145 mg every 4 weeks for 12 weeks
- AEGR-733 5 mg + Ezetimibe 10 mg: Oral lomitapide 5 mg + ezetimibe 10 mg every 4 weeks for 12 weeks
Period: Overall Study
Arm/Group | Placebo | AEGR-733 2.5 mg | AEGR-733 5 mg | AEGR-733 7.5 mg | AEGR-733 10 mg | AEGR-733 5 mg + Atorvastatin 20 mg | AEGR-733 5 mg + Fenofibrate 145 mg | AEGR-733 5 mg + Ezetimibe 10 mg
Started | 33 | 34 | 34 | 34 | 35 | 28 | 33 | 29
Completed | 31 | 25 | 24 | 29 | 21 | 23 | 28 | 25
Not Completed | 2 | 9 | 10 | 5 | 14 | 5 | 5 | 4
Not completed — Adverse Event | 1 | 7 | 8 | 5 | 11 | 4 | 4 | 2
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 2 | 0 | 3 | 1 | 0 | 2
Not completed — Inclusion/exclusion criteria not met | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | AEGR-733 2.5 mg | AEGR-733 5 mg | AEGR-733 7.5 mg | AEGR-733 10 mg | AEGR-733 5 mg + Atorvastatin 20 mg | AEGR-733 5 mg + Fenofibrate 145 mg | AEGR-733 5 mg + Ezetimibe 10 mg | Total
Number analyzed (Participants) | 33 | 34 | 34 | 34 | 35 | 28 | 33 | 29 | 260
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.8 (12.53) | 51.5 (12.99) | 48.6 (11.3) | 49.0 (10.24) | 52.9 (11.97) | 53.9 (8.92) | 54.0 (11.95) | 52.7 (9.36) | 51.3 (11.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 18 | 16 | 17 | 20 | 17 | 17 | 12 | 136
  Male | 14 | 16 | 18 | 17 | 15 | 11 | 16 | 17 | 124
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 9 | 8 | 9 | 8 | 4 | 7 | 5 | 55
  White | 24 | 21 | 24 | 23 | 22 | 22 | 24 | 22 | 182
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 4 | 2 | 1 | 5 | 2 | 1 | 2 | 20
Region of Enrollment [Number; unit: participants]
  United States | 33 | 34 | 34 | 34 | 35 | 28 | 33 | 29 | 260

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change From Baseline in Percent Hepatic Fat
Description: Absolute change from Baseline in percent hepatic fat
Time Frame: Baseline and 12 weeks on study drug
Population: ITT
Measure: Mean (Standard Deviation); unit: Percent of Hepatic Fat
Arm/Group | Placebo | AEGR-733 5 mg
Number analyzed (Participants) | 31 | 24
Percent of Hepatic Fat | 0.03 (1.814) | 4.72 (6.297)
Statistical Analysis 1: Comparison: Placebo vs AEGR-733 5 mg; One-way analysis of variance (ANOVA) to compare the absolute change from baseline to Week 12 in percent hepatic fat between AEGR-755 5 mg and placebo; Test type: Superiority or Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 4.68, 95% CI 2-sided [2.30 to 7.07]

2. Secondary Outcome: Absolute Change From Baseline in Percent Hepatic Fat
Description: Absolute change from Baseline in percent hepatic fat
Time Frame: Baseline and 12 weeks on study drug
Population: ITT
Measure: Mean (Standard Deviation); unit: Percent of Hepatic Fat
Arm/Group | Placebo | AEGR-733 2.5 mg | AEGR-733 5 mg | AEGR-733 7.5 mg | AEGR-733 10 mg | AEGR-733 5 mg + Atorvastatin 20 mg | AEGR-733 5 mg + Fenofibrate 145 mg | AEGR-733 5 mg + Ezetimibe 10 mg
Number analyzed (Participants) | 31 | 27 | 24 | 27 | 20 | 23 | 26 | 26
Percent of Hepatic Fat | 0.03 (1.814) | 4.95 (7.122) | 4.72 (6.297) | 3.94 (5.763) | 7.86 (9.515) | 3.68 (5.365) | 7.70 (9.390) | 7.55 (6.230)
Statistical Analysis 1: Comparison: Placebo vs AEGR-733 2.5 mg; One-way ANOVA to compare the absolute change from baseline to Week 12 in percent hepatic fat between active treatment groups and placebo; Test type: Superiority or Other; p < 0.001, ANOVA — (All comparisons); Mean Difference (Final Values) = 4.92, 95% CI 2-sided [2.27 to 7.57]
Statistical Analysis 2: Comparison: Placebo vs AEGR-733 5 mg; Test type: Superiority or Other; p < 0.001, ANOVA — (All comparisons); Mean Difference (Final Values) = 4.68, 95% CI 2-sided [2.30 to 7.07]
Statistical Analysis 3: Comparison: Placebo vs AEGR-733 7.5 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, ANOVA — (All comparisons); Mean Difference (Final Values) = 3.91, 95% CI 2-sided [1.73 to 6.10]
Statistical Analysis 4: Comparison: Placebo vs AEGR-733 10 mg; Test type: Superiority or Other; p < 0.001, ANOVA — (All comparisons); Mean Difference (Final Values) = 7.82, 95% CI 2-sided [4.31 to 11.33]
Statistical Analysis 5: Comparison: Placebo vs AEGR-733 5 mg + Atorvastatin 20 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, ANOVA — (All comparisons); Mean Difference (Final Values) = 3.65, 95% CI 2-sided [1.58 to 5.72]
Statistical Analysis 6: Comparison: Placebo vs AEGR-733 5 mg + Fenofibrate 145 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, ANOVA — (All comparisons); Mean Difference (Final Values) = 7.66, 95% CI 2-sided [4.22 to 11.11]
Statistical Analysis 7: Comparison: Placebo vs AEGR-733 5 mg + Ezetimibe 10 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, ANOVA — (All comparisons); Mean Difference (Final Values) = 7.51, 95% CI 2-sided [5.16 to 9.86]

ADVERSE EVENTS:
Time Frame: From 10 days before the first dose to 30 days post last dose.
Arm/Group | Placebo | AEGR-733 2.5 mg | AEGR-733 5 mg | AEGR-733 7.5 mg | AEGR-733 10 mg | AEGR-733 5 mg + Atorvastatin 20 mg | AEGR-733 5 mg + Fenofibrate 145 mg | AEGR-733 5 mg + Ezetimibe 10 mg
Serious Adverse Events (participants affected / at risk) | 0/33 | 1/34 | 0/34 | 0/34 | 2/35 | 0/28 | 0/33 | 0/29
Other Adverse Events (participants affected / at risk) | 20/33 | 31/34 | 30/34 | 29/34 | 32/35 | 24/28 | 29/33 | 25/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=33) | AEGR-733 2.5 mg (N=34) | AEGR-733 5 mg (N=34) | AEGR-733 7.5 mg (N=34) | AEGR-733 10 mg (N=35) | AEGR-733 5 mg + Atorvastatin 20 mg (N=28) | AEGR-733 5 mg + Fenofibrate 145 mg (N=33) | AEGR-733 5 mg + Ezetimibe 10 mg (N=29)
Chest Pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Inflammatory Bowel Disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ankle Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=33) | AEGR-733 2.5 mg (N=34) | AEGR-733 5 mg (N=34) | AEGR-733 7.5 mg (N=34) | AEGR-733 10 mg (N=35) | AEGR-733 5 mg + Atorvastatin 20 mg (N=28) | AEGR-733 5 mg + Fenofibrate 145 mg (N=33) | AEGR-733 5 mg + Ezetimibe 10 mg (N=29)
Diarrhoea (Gastrointestinal disorders) | 4 | 16 | 15 | 16 | 23 | 14 | 15 | 19
Nausea (Gastrointestinal disorders) | 1 | 2 | 8 | 8 | 13 | 5 | 8 | 5
Headache (Nervous system disorders) | 4 | 2 | 6 | 8 | 1 | 3 | 4 | 4
Flatulence (Gastrointestinal disorders) | 2 | 6 | 3 | 1 | 2 | 5 | 1 | 6
Fatigue (General disorders) | 2 | 3 | 5 | 3 | 3 | 1 | 3 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 2 | 2 | 2 | 5 | 4 | 2 | 2 | 1
Abdominal Distension (Gastrointestinal disorders) | 2 | 2 | 3 | 4 | 1 | 2 | 2 | 2
Vomiting (Gastrointestinal disorders) | 1 | 2 | 3 | 1 | 4 | 2 | 5 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 4 | 1 | 1 | 2 | 2 | 2 | 4
Constipation (Gastrointestinal disorders) | 3 | 0 | 0 | 1 | 0 | 2 | 4 | 2
Abdominal Pain (Gastrointestinal disorders) | 2 | 2 | 3 | 1 | 3 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 3 | 0 | 2 | 1 | 0 | 1 | 0 | 4
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2 | 2 | 1 | 0 | 1 | 2
Alanine Aminotransferase Increased (Investigations) | 0 | 3 | 2 | 1 | 1 | 0 | 4 | 0
Aspartate Aminotransferase Increased (Investigations) | 0 | 2 | 1 | 1 | 1 | 0 | 4 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 1 | 0 | 2 | 0 | 0 | 4 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1 | 0 | 1 | 1 | 3 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 1 | 2 | 0 | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 1 | 0 | 1 | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4 | 0 | 1 | 0 | 0 | 2
Dizziness (Nervous system disorders) | 1 | 1 | 2 | 0 | 1 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 2
Seasonal Allergy (Immune system disorders) | 0 | 0 | 1 | 2 | 1 | 0 | 2 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 2 | 2 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0 | 1 | 2 | 2 | 0
White Blood Cell Count Decreased (Investigations) | 1 | 2 | 1 | 0 | 0 | 0 | 1 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1
Protein Urine (Investigations) | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Influenza Like Illness (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Gastrointestinal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Eruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
C-reactive Protein (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI can publish after sponsor reviews the proposed publication. PI must give sponsor at least 60 days to review before publication. PI needs to obtain sponsor's prior written consent to publish confidential information, which shall not be unreasonably withheld or delayed. The PI shall, upon request of sponsor, delete any confidential information which would prejudice the securing of adequate intellectual property protection from the publication.